CLINICAL TRIAL: NCT05923281
Title: A Phase III Confirmatory Study of K-877 (Pemafibrate) in Patients With Hypercholesterolemia and Statin Intolerance-Multicenter, Placebo Controlled, Randomized, Double Blind, Parallel Group Controlled Trial in Patients With Statin Intolerant Hypercholesterolemia-
Brief Title: A Phase III Confirmatory Study of K-877 (Pemafibrate) in Patients With Hypercholesterolemia and Statin Intolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-877-ER-04
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): K-877 0.2 mg/day
  Interventions: Drug: K-877 0.2 mg/day (once daily)
- Treatment B (Experimental): K-877 0.4 mg/day
  Interventions: Drug: K-877 0.4 mg/day (once daily)
- Control A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (once daily)

INTERVENTIONS:
Drug: K-877 0.2 mg/day (once daily) — K-877 0.2mg tablet
  Other Names: Pemafibrate 0.2mg/day (once daily)
  Arms: Treatment A
Drug: K-877 0.4 mg/day (once daily) — K-877 0.2mg tablet
  Other Names: Pemafibrate 0.4mg/day (once daily)
  Arms: Treatment B
Drug: Placebo (once daily) — Placebo tablet
  Arms: Control A

SUMMARY:
To investigate the efficacy and safety of K-877 Extended Release 0.2 mg/day or 0.4 mg/day for 12 weeks in patients with Statin Intolerant* Hypercholesterolemia,using placebo as a controll.

*Statin Intolerant: Adverse events associated with statin use that cause unacceptable disturbances in the user's daily life, resulting in drug discontinuation or dose reduction.

ELIGIBILITY:
Inclusion Criteria: The person who meet all the following criteria the object to the clinical trial

1. Patients had to be age 18 years or older at written informed consent
2. Patients with statin intolerant hypercholesterolemia
3. Patients who have laboratory records with fasting serum TG <= 150 mg/dL (<=175 mg/dL when not fasting) within 6 months prior to consent.
4. Patients with the fasting serum TG <= 150 mg/dL at screening
5. Patients who have received dietary or exercise guidance from 12 weeks or more prior to Screening
6. Patients who apply any of the following risk category with LDL-C level (Friedewald formula) based on JAS2022 at screening

   * Low risk for primary prevention: LDL-C >=160 mg/dL
   * Intermediate risk for primary prevention: LDL-C >=140 mg/dL
   * High risk for primary prevention: LDL-C>=120 mg/dL
   * Secondary prevention: LDL-C>=120 mg/dL

Exclusion Criteria: The person who meet any of the following criteria will be excluded from the study.

1. Patients who require administration of prohibited drugs during the clinical trial period after written informed consent
2. Patients with type 1 diabetes and uncontrolled diabetes [HbA1c(NGSP) >= 10.0 % at Screening]
3. Patients with uncontrolled thyroid disease
4. Patients with undergoing LDL apheresis
5. Patients with cirrhosis or those with biliary obstruction
6. Patients with familial hypercholesterolemia (homozygotes)
7. Patients with uncontrolled hypertension (SBP >= 160 mmHg or DBP >= 100 mmHg) at Screening
8. Patients with an AST or ALT three times the upper limit at Screening
9. Patients with an CK four times the upper limit at Screening
10. Patients with any of the following criteria within 3 months before obtaining informed consent: myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass surgery, stroke, transient ischemic attack, symptomatic carotid artery stenosis, symptomatic peripheral arterial disease, abdominal aortic aneurysm, uncontrolled severe arrhythmia and decompensated heart failure
11. Patients who plan to undergo PCI, CABG, carotid artery or peripheral revascularization
12. Patients with heart failure class III or higher according to NYHA cardiac function classification
13. Patients with malignant tumor or those who are judged to have a high risk of recurrence
14. Patients with a history of myopathy or rhabdomyolysis due to K-877 (pemafibrate)
15. Patients with a history of hypersensitivity due to K-877 (pemafibrate)
16. Patients with a history of serious drug allergies (anaphylactic shock, etc.)
17. Pregnant women, lactating women, women planning to become pregnant or lactating during the study period, or pregnant women*2 who do not use specific contraceptive methods*1
18. Patients who have collected 400 mL or more of whole blood within 16 weeks, or 200 mL or more of whole blood within 4 weeks, or blood samples (plasma and platelet components) within 2 weeks before Screening
19. Patients with alcoholics or drug addicts
20. Patients who participated in other clinical trials of a drug with new active ingredients within 16 weeks or a drug with an approved active ingredients within 12 weeks prior to administration and received an investigational drug other than placebo,or those who will participate in other clinical trials at the same time as the clinical trial
21. Patients who have been determined inappropriate by the investigator, etc

    * 1 Acceptable contraceptive methods: oral, implantable/injectable contraceptive hormones, mechanical products [intrauterine devices (IUDs) ,etc] or barrier methods with spermicides (pessaries, condoms, cervical caps, etc)
    * 2 Woman of childbearing potential refers to a woman who is physiologically capable of becoming pregnant with a male partner who has not undergone contraception. However, it does not apply if the investigator confirms that any of the following criteria is met.

      * Patients with hysterectomy or tubal ligation before informed consent
      * Post-menopausal women (those who who have passed more than 1 year since their last menstrual period without other medical reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C (formula F). | 4, 8, and 12 weeks after administration
  Percent change = (measured value at each time point - baseline value) / baseline value

SECONDARY OUTCOMES:
Efficacy: % change from baseline in fasting serum LDL-C (mg/dL)(Direct) | 4, 8, and 12 week after administration
Efficacy: % change from baseline in fasting serum HDL-C (mg/dL) | 4, 8, and 12 week after administration
Efficacy: % change from baseline in fasting serum non HDL-C (mg/dL) | 4, 8, and 12 week after administration
Efficacy: % change from baseline in fasting serum TG (mg/dL) | 4, 8, and 12 week after administration
Efficacy: % change from baseline in fasting serum LDL-C（formula F）/HDL-C | 4, 8, and 12 week after administration
Efficacy: % change from baseline in fasting serum non HDL-C/HDL-C | 4, 8, and 12 week after administration

CONTACTS AND LOCATIONS:
Locations (22):
- Japan (22):
  - Nakayama Clinic, Aichi
  - Kohnodai Hospital, National Center for Global Health and Medicine, Chiba
  - Tashiro Endocrinology Clinic, Fukuoka
  - Central Japan International Medical Center, Gifu
  - NTT Medical Center Sapporo, Hokkaido
  - Tsukuba Medical Center Foundation Tsukuba Medical Center Hospital, Ibaraki
  - Yokohama Minami Kyosai Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Medical Corporation LONGWOOD Maeda Clinic, Osaka
  - OCROM Clinic, Osaka
  - Rinku General Medical Center, Osaka
  - Koshigaya Municipal Hospital, Saitama
  - Saitama Medical University Hospital, Saitama
  - Affiliated CENTRAL CLINIC of Higashiyamato Hospital, Tokyo
  - Fukuwa Clinic, Tokyo
  - Juntendo University Hospital, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Tokyo
  - Mishuku Hospital, Tokyo
  - Seiwa Clinic, Tokyo
  - ToCROM Clinic, Tokyo
  - Tokyo Heart Summit Tokyo Heart Rhythm Hospital, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo